| Official Protocol Title: | RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY TO ASSESS CARDIOVASCULAR OUTCOMES FOLLOWING TREATMENT WITH ERTUGLIFLOZIN (MK-8835/PF-04971729) IN SUBJECTS WITH TYPE 2 DIABETES MELLITUS AND ESTABLISHED VASCULAR DISEASE, THE VERTIS CV STUDY |
|---|---|
| NCT number: | NCT01986881 |
| <b>Document Date:</b> | 20-Mar-2020 |

Statistical Analysis Plan for secondary analyses of heart failure and related outcomes in the VERTIS CV trial (Trial B1521021)
Version 4

Final version - March 20th, 2020

Final formatting - March 24th, 2020

Primary Author:

Input from SAC members/co-authors

**Sponsor Co-authors:** 

VERTIS CV is a multinational, placebo-controlled, double-blind, randomized, parallel-group Phase III trial to assess the impact of ertugliflozin therapy on cardiovascular (CV) outcomes in a population with type 2 diabetes mellitus (T2DM) and a history of atherosclerotic cardiovascular disease (ASCVD).

Here we describe the statistical considerations for additional exploratory analyses to further investigate the impact of ertugliflozin on heart failure (HF)-related outcomes to complement the primary assessment of HHF/CVD death in the primary statistical hierarchy and secondary outcomes of HHF. This document is a supplement to the HF hospitalization and related analyses in the protocol and the primary SAP, and is intended to prospectively specify a series of 'hypothesis-generating analyses'. Additional exploratory analyses may be conducted in the future based upon the results of the pre-specified analyses of HF related outcomes.

### 1. Background and Rationale

Time to composite of hospitalization for heart failure (HHF) and CV death defined as time from randomization to a confirmed event of hospitalization for HF or CV related death (i.e., an event meeting adjudication criteria) is a pre-specified VERTIS CV outcome included in the primary statistical analysis hierarchy. All reported hospital admissions for HF, including first and any recurrent events, will be CEC adjudicated. In addition HHF alone (time to first) is one of the secondary outcomes.

CEC-adjudicated events of hospitalization for HF are recognized as a standard component in HF development programs (either as an efficacy or a safety parameter, according to the specific program goals). Assessed in a controlled clinical study, the frequency of HF hospitalizations is expected to be driven by acute decompensations and correlate with general HF disease progression in a given cohort. However, although generally accepted by the clinical community, it is recognized that time to first event outcome has a number of limitations. For example, it does not incorporate analysis of recurrent events or does not consider results based on the presence or absence of HF at baseline including type of heart failure (HFrEF; HFpEF). Given the demonstrated benefit for the SGLT2 class on HHF and composite HHF/CV death diabetic population as well as recent publication demonstrating reduction in CV events in subjects with HFrEF without diabetes (DAPA HF reference) there is significant scientific interest in CV outcomes in subjects with different types of HF. Significant proportion of subjects in VERTIS CV had heart failure prior to study enrollment therefore additional prespecified analyses will be conducted to explore effects of ertugliflozin on reduction of HF related CV events/CV death.

#### **Baseline characteristics:**


Summary of baseline population characteristics will be presented in a tabular form by a) by presence or absence of prior HF at baseline and-randomized treatment assignment; and b) in subset of patients with prior history of HF by EF: rEF, pEF, and unknown EF and treatment assignment; and c)independent of prior HF status, stratified by EF: rEF; pEF; and Unknown EF and treatment assignment. Format used will be similar to that in <a href="Example">Example</a> of potential display below (CARMELINA paper Table#1)

Overall study population (N = 8246; reference to primary publication)

- a) Comparison of baseline characteristics, all ertu versus placebo based on baseline history of heart failure = Yes/No
  - b) Summary of baseline characteristics among those with prior HF by type of heart failure (same characteristics as above; table would have 3 column headings (HFrEF; HFpEF; HFunkEF + heart failure history = yes but with no baseline EF available)
  - c) overall study cohort by EF: rEF, pEF, and unknown EF.

| ble 1. Baseline Characteristics of Participan | | | 1 | | 1 |
|---|---|---|---|---|---|
| Characteristic | Participants Wi<br>Linagliptin | th HF at Baseline<br>Placebo | Participants With<br>Linagliptin | out HF at Baseline<br>Placebo | Total CARMELINA<br>Population |
| N (%) | 952 (100) | 921 (100) | 2542 (100) | 2564 (100) | 6979 (100) |
| Age, y | 66.5 (8.64) | 65.8 (8.95) | 65.9 (9.2) | 65.6 (9.2) | 65.9 (9.10) |
| Male, n (%) | 561 (58.9) | 581 (63.1) | 1587 (62.4) | 1661 (64.8) | 4390 (62.9) |
| Race, n (%) | | | | 7.5.5.5.5.5.5.5.5.5.5.5.5.5.5.5.5.5.5.5 | |
| White | 845 (88.8) | 813 (88.3) | 1982 (78.0) | 1956 (76.3) | 5596 (80.2) |
| Asian | 38 (4.0) | 26 (2.8) | 269 (10.6) | 307 (12.0) | 640 (9.2) |
| Black/African American | 43 (4.5) | 57 (6.2) | 151 (5.9) | 160 (6.2) | 411 (5.9) |
| Other* | 26 (2.7) | 25 (2.7) | 140 (5.5) | 141 (5.5) | 332 (4.8) |
| Region, n (%) | | | | | |
| Europe (including South Africa) | 589 (61.9) | 572 (62.1) | 884 (34.8) | 889 (34.7) | 2934 (42.0) |
| Latin America | 187 (19.6) | 192 (20.8) | 969 (38.1) | 962 (37.5) | 2310 (33.1) |
| North America | 142 (14.9) | 136 (14.8) | 451 (17.7) | 451 (17.6) | 1180 (16.9) |
| Asia | 34 (3.6) | 21 (2.3) | 238 (9.4) | 262 (10.2) | 555 (8.0) |
| Smoking status, n (%) | | | | | |
| Never smoker | 553 (58.1) | 539 (58.5) | 1344 (52.9) | 1317 (51.4) | 3753 (53.8) |
| Ex-smoker | 310 (32.6) | 300 (32.6) | 921 (36.2) | 976 (38.1) | 2507 (35.9) |
| Current smoker | 88 (9.2) | 81 (8.8) | 274 (10.8) | 269 (10.5) | 712 (10.2) |
| Missing | t (0.1) | 1 (0.1) | 3 (0.1) | 2 (0.1) | 7 (0.1) |
| History of heart failure, n (%) | 952 (100) | 921 (100) | 0 (0) | 0 (0) | 1873 (26.8) |
| ischemic heart disease, n (%) | 745 (78.3) | 760 (82.5) | 1284 (50.5) | 1292 (50.4) | 4081 (58.5) |
| History of hypertension, n (%) | 884 (92.9) | 855 (92.8) | 2287 (90.0) | 2323 (90.6) | 6349 (91.0) |
| Atrial fibrillation, n (%) | 171 (18.0) | 171 (18,6) | 148 (5.8) | 183 (7.1) | 673 (9.6) |
| eGFR (MDRD), mL/mlrv1.73 m <sup>2</sup> | 55.8 (24.3) | 55.1 (24.7) | 54.2 (25.4) | 54.3 (25.0) | 54.6 (25.0) |
| eGFR (MDRD), n (%) | | | | | |
| ≥60 mL/mln/1,73 m <sup>2</sup> | 367 (38.6) | 367 (39.8) | 927 (36.5) | 970 (37.8) | 2631 (37.7) |
| ≥45 to <60 mL/min/1.73 m <sup>2</sup> | 208 (21.8) | 166 (18.0) | 482 (19.0) | 492 (19.2) | 1348 (19.3) |
| ≥30 to <45 mL/min/1.73 m <sup>2</sup> | 263 (27.6) | 249 (27.0) | 731 (28.8) | 695 (27.1) | 1938 (27.8) |
| <30 mL/mir/1.73 m <sup>2</sup> | 114 (12.0) | 139 (15.1) | 402 (15.8) | 407 (15.9) | 1062 (15.2) |
| UACR, mg/g, median (25th-75th percentile) | 139 (36–589) | 158 (46-727) | 173 (47–753) | 163 (43-758) | 162 (44-728) |
| UACR, n (%)† | | | | | |
| <30 mg/g | 215 (22.6) | 184 (20.0) | 481 (18.9) | 512 (20.0) | 1392 (19.9) |
| 30-300 mg/g | 397 (41.7) | 389 (42.2) | 1066 (41.9) | 1042 (40.6) | 2894 (41.5) |
| >300 mg/g | 340 (35.7) | 348 (37.8) | 993 (39.1) | 1009 (39.4) | 2690 (38.5) |

McGuire et al

#### 2. Analysis of time to first event of HF hospitalizations (HHF) and of HHF/CV Death composite

#### The VERTIS protocol and primary SAP already include (Tables and KM will be available):

- a) Secondary hypothesis superiority testing time to the first composite of HHF/CV death as prespecified efficacy outcome, which will be analyzed both in the intention-to-treat (CV ITT; primary analysis strategy) and the on treatment analysis (CV FAS with +14 and +30 days censoring window) utilizing Cox Proportional Hazard (CPH) statistical method.
- b) Secondary outcome of time to first Hospitalization for HF utilizing CPH model (CVITT and on treatment CV FAS + 14 days)
- c) NEW: KM-individual treatment groups (5 mg, 15 mg) for HHF will be generated (KM individual treatment groups for the composite already exists)

#### Additional proposed analysis will include (Tables and KM curves):

- I. Time to event analyses using Cox proportional hazards models will be performed for these assessments, using the Fine and Gray method to account for competing risk of non-CV mortality in analyses of the HHF/CV Death composite outcome (CV ITT) and HHF (CV ITT). Exposure times of all patients will be censored at the date they were last known to be free of all components of the individual and composite outcomes analyzed.
- II. A supportive analysis for the composite HHF/CV Death and HHF will be performed (CPH, CV ITT) in the subsets of patients with history of HF at baseline (1900/8238; 23.1%), and in those without prior HF. The time to first confirmed event will be modeled univariably with treatment, and also in multivariable analyses including region and baseline type of ASCVD status as ASCVD risk factors. Baseline CVD status /risk factors will include 5 different model terms:
  - o CAD,
  - o cerebrovascular disease,
  - o PVD.
  - o prior MI,
  - o prior stroke

In addition, univariablee analyses CPH (CV ITT) with factor for HF at baseline will be conducted for:

- MACE;
- HHF/CV Death;
- CV death;
- HHF
- All-cause death

#### 3. Total events (composite of HF hospitalization or CV death)

The classical analysis of time to first event has the disadvantage of excluding all events that occur subsequent to the first. In order to gain maximal information from the study, it is important to consider events that occur after a first non-fatal event has occurred.


I. Analyses will be performed to explore the effect of ertugliflozin on total events including the first and subsequent events for HHF and HHF/CV Death outcomes. Anderson-Gill method will be used as the primary analysis method (CV ITT) to analyze multiple occurrences of these outcomes (1 event, 2 events, ≥3 events), with treatment as an explanatory factor, region as a stratification factor, and history of HF and CVD status at baseline as other factors. CVD status will include CAD, cerebrovascular disease, PVD, prior MI, and prior stroke. A point estimate and two sided 95% confidence interval for the hazard ratio and the resulting p value will be reported. Descriptive statistics will also be reported for recurrent events, displaying the number of patients with 1, 2, and ≥3 events) by treatment group.

Alternative methods for analyses of first + recurrent events, including Wei-Lin-Weisfeld (WLW) method, negative binomial regression and frailty models will not be used in initial analysis but will be provided as sensitivity analyses if requested by the peer review process.

#### 4. Subgroup analyses (table /forest plots).

Analyses of time to first event of HHF and of HHF/CV death (CV ITT), pooled doses, stratified by the following baseline characteristics will be included, using formal test of heterogeneity of the treatment effect among these subgroups:

- Median split for age
- Sex
- Race
- Ethnicity
- Region
- Median split BMI
- Median split for diabetes duration
- Baseline  $< 8.5, \ge 8.5\%$  HbA1c
- Baseline UACR (<30; 30-300; and >300)
- Baseline ACEI/ARB
- Baseline MRA use
- Baseline beta blocker use
- Baseline loop diuretic use
- Baseline insulin use
- Baseline metformin use
- Prior HF
- Ejection Fraction (<40%; 40-50%; >50%; unknown EF)
- Prior MI (Yes/No)
- CAD (Yes/No)
- Atrial fibrillation
- Hypertension
- Baseline eGFR (<45, 45<60, 60 <90, and >90) and dichotomously by eGFR <60: Y/N

- 5. Additional analyses of time to first primary and key secondary outcomes (CV ITT population) by EF (< 45%; ≥45%; unknown):
  - a) among those with HF at baseline; and
  - b) in the overall population regardless of HF history at baseline:

Forest plots will be available for primary and key efficacy outcomes based on presence or absence of prior HF at baseline.

#### **Additional exploratory analyses:**

I) Time to first primary and key secondary outcomes stratified by EF (CV ITT population)

Analyses of the primary and key efficacy outcomes will be presented based on type of HF in patients with HF at baseline, and in the entire population regardless of HF presence at baseline (EF cut off <45):

- a) 6 groups:
  - rEF and HF+
  - rEF and HF-
  - pEF and HF+
  - pEF and HF-
  - unk EF and HF+
  - unk EF and HF-
- b) Entire study population analyses based on EF alone regardless of HF status:
  - rEF
  - pEF
  - unkEF

## Data will be produced for:

- MACE;
- CV/HHF composite;
- CV death;
- HHF;
- All-cause death;
- HHF or CV death (all first + recurrent)
- HHF or all-cause death (all first + recurrent)


# II) Descriptive summary of readmissions and death among subjects who experienced at least one HHF (CV ITT), Example table 14.2.20 below:

- Descriptive summary of readmissions and deaths among subjects w/ at least one HHF event in study
- Same as previous but broken down by prior HF at baseline
- Same as previous but broken down by EF (45) at baseline
- Same as previous but broken down by HF/EF category at baseline

### 6. Absolute difference NNT table for the following outcomes:

- MACE
- CV Death
- All cause mortality
- HHF
- HHF or CV Death

### 7. High level summary of key safety findings:

CV SOC table / High Level Group Term or PT (MeDRA dictionary SOC only) (AFib , CHF AEs etc - expecting less AEs in active arm.

## **APPENDIX 1:**

8. Additional future analyses for consideration beyond the initial publication at ESC (perhaps for AHA 2020 or ACC 2021):

I. Benchmark analysis similar to what was presented in prior publications.



II. Time to onset of effect similar as presented for DAPA HF, AHA meeting 2019.



## III. Heart failure risk stratification analysis - paper similar to Berg et al.

0

## Circulation

## ORIGINAL RESEARCH ARTICLE

Heart Failure Risk Stratification and Efficacy of Sodium-Glucose Cotransporter-2 Inhibitors in Patients With Type 2 Diabetes Mellitus

#### Berg et al

#### Table 2. TRS-HF<sub>DM</sub> In the Derivation Cohort

| Risk Indicator | Adjusted HR (95% CI) | P Value | Points |
|---|---|---|---|
| Prior heart failure | 4,22 (3.18-5.59) | <0.001 | 2 |
| Atrial fibrillation | 2.26 (1.62-3.14) | <0.001 | 1 |
| Coronary artery disease | 2.06 (1.45-2.93) | <0.001 | 1 |
| eGFR <60 mL-min <sup>-1</sup> -1.73 m <sup>-2</sup> | 1.85 (1.40-2.46) | <0.001 | 1 |
| Urine albumin-to-creatinine ra | tio | | |
| >300 mg/g | 4.50 (3.18-6.36) | <0.001 | 2 |
| 30-300 mg/g | 2.08 (1.50-2.87) | <0.001 | 1 |

eGFR <60 mL·min<sup>-1</sup>·1.73 m<sup>-2</sup> represents chronic kidney disease. Urine albumin-to-creatinine ratio 30–300 mg/g represents moderately increased albuminuria, whereas >300 mg/g represents severely increased albuminuria. eGFR indicates estimated glomerular filtration rate; HR, hazard ratio; TIMI, Thrombolysis in Myocardial infarction; and TRS-HF<sub>DM</sub>, TIMI Rtsk Score for Heart Failure in Diabetes.

Berg et al Heart Failure Risk Stratification in Diabetes



Figure 2. Treatment effect of dapagliflozin by baseline risk of hospitalization for heart failure. Although relative risk reductions were similar across risk score categories, absolute reductions in Kaplan-Meier estimates of hospitalization for heart failure risk at 4 years were greater in those at higher baseline risk (yi-3.24; 1-sided Pfor trend=0,04). ARR Indicates absolute risk reduction; HR, hazard ratio; and NNT, number needed to treat.

### IV. Future biomarker analyses in 2021 – biomarkers TBD

APPENDIX 2: Below section includes only key reference points with regards to primary SAP and data collection (background material):

Statistical considerations: Existing key analyses primary SAP:

#### Stage 2 Analyses

| Eudpoint | Analysis Set | Statistical Method | Ascertainment<br>Window (Days) | Description |
|---|---|---|---|---|
| MACE | CVFAS | СРН | 365 | Primary NI analysis |
| | CVITT | | No limit | On-study analysis |
| | CVFAS | | 14 | On-treatment analysis |
| | | | 30 | On-treatment analysis |
| | | Min Risk | 365 | Sensitivity analysis |
| CV death/HHF | CVITT | CPH | No limit | Secondary superiority analysis |
| | CVFAS | | 14 | On-treatment analysis |
| | 1 | | 30 | On-treatment analysis |
| CV death | CVITI | CPH | No limit | Secondary superiority analysis |
| | CVFAS | 1000 | 14 | On-treatment analysis |
| | | | 30 | On-treatment analysis |
| Renal composite | CVITT | СРН | No limit | Secondary superiority analysis |
| | CVFAS | | 14 | On-treatment analysis |
| | | | 30 | On-treatment analysis |
| MACE plus | CVITT | СРН | No limit | Secondary analysis |
| | CV FAS | | 14 | On-treatment analysis |
| FNF MI | CVITT | CPH | No limit | Secondary analysis |
| | CVFAS | | 14 | On-treatment analysis |
| FNF stroke | CVITT | CPH | No limit | Secondary analysis |
| | CVFAS | | 14 | On-treatment analysis |
| Hospitalization for HF | CVITT | CPH | No limit | Secondary analysis |
| North Control of the | CVFAS | | 14 | On-treatment analysis |
| All-cause mortality | CVITT | CPH | No limit | Secondary analysis |
| | CVFAS | | 14 | On-treatment analysis |
| Total MACE | CVITT | Andersen-Gill | No limit | Exploratory analysis |
| Total CV death/HHF | CVITT | Andersen-Gill | No limit | Exploratory analysis |

MACE-Major Adverse Cardiovascular Event: FNF=Fatal or Non-Fatal. MI=Myocardial Infarction; UA=unstable angina; HF=Heart Failure; NI = Non-Inferiority

#### **Subgroup analysis primary SAP:**

For Stage 2, analyses of MACE and the secondary CV endpoints included in the formal testing sequence will be performed in subgroups based on region, gender, age (<65 and  $\geq$ 65 years), race, ethnicity, category of chronic kidney disease (CKD; based on baseline eGFR: <60, 60 to <90, and  $\geq$ 90 mL/min/1.73 m²), history of heart failure, baseline HbA1c (<8.5 and  $\geq$ 8.5%), baseline BMI (<30 and  $\geq$ 30 kg/m²), and use of the following concomitant medications at baseline: statins, ezetimibe, ASA/anti-platelets, diuretics, beta blockers, calcium channel blockers, mineralocorticoid receptor antagonists, renin-

PFIZER CONFIDENTIAL Page 24

Protocol MK-8835-004-01/B1521021

Statistical Analysis Plan

angiotensin-aldosterone system (RAAS) blockers, insulin, DPP-IV inhibitors, metformin, sulfonylureas, and GLP-1 agonists. Selected subgroups (to be specified in the list of tables) will also be analyzed for the renal composite endpoint. These subgroup analyses will be considered exploratory and will not be adjusted for multiple comparisons. The same model used for the primary analysis will be run within each subgroup. The data will also be summarized descriptively by treatment group within each subgroup.

In order to provide model-based point and interval estimates of the hazard ratios for MACE and the endpoints in the formal testing sequence for each dose of ertugliflozin (5 mg and 15 mg), an analysis of Study B1521021 will be conducted using the individual dose groups.

For Stage 2, a summary of the sub-group of subjects experiencing at least one adjudicated and confirmed hospitalization for heart failure will be produced in order to evaluate these subjects for all-cause and CV mortality (including the adjudicated causes of death) and seed white for the produced for heart failure.

## **Key data collection reference points:**


#### Collection of Background CV conditions at baseline:

Associated Vascular Diagnosis (AVD) CRF page: Collected on all subjects with instructions to mark conditions if they met protocol Inclusion #4 criteria:

| Coronary Artery<br>Disease | ◆ Select the appropriate response ◆ Absent ◆ Present |
|---|---|
| Cerebrovascular<br>Disorder | ◆ Select the appropriate response ◆ Absent ◆ Present |
| Peripheral Arterial<br>Disease | ◆ Select the appropriate response |

#### **Inclusion #4**

- Subjects must have evidence or a history of atherosclerosis involving the coronary, cerebral or peripheral vascular systems as follows (must have at least one of the following a-d):
  - a. <u>Coronary artery disease</u> as indicated by a history of presumed spontaneous myocardial infarction (hospitalized with final diagnosis of myocardial infarction, excluding peri-procedural or definite secondary myocardial infarction [eg, due to profound anemia or hypertensive emergency, troponin increase in sepsis] in which the most recent event occurred at least 3 months (90 days) prior to the Screening visit (V1); OR
  - b. <u>Coronary artery disease</u> as indicated by a history of coronary revascularization through either a Percutaneous Coronary Intervention (PCI) at least 3 months (90 days) prior to the Screening visit (V1) or Coronary Artery Bypass Graft (CABG) at least 3 months (90 days) prior to the Screening visit (V1); OR
  - c. <u>Ischemic (presumed thrombotic) cerebrovascular disease</u> as indicated by a history of ischemic stroke (hospitalized with a final diagnosis of non-hemorrhagic stroke [includes completion of a standard evaluation for stroke in an acute care facility or stroke clinic without hospital admission] with the most recent event occurring at least 3 months (90 days) prior to the Screening visit (V1) or a history of carotid revascularization at least 3 months (90 days) prior to the Screening visit (V1); OR
  - d. Peripheral arterial disease as indicated by:
    - 1. Angiographically-documented peripheral vascular disease; or
    - Resting ankle/brachial index (ABI) of <0.85 (measured by a certified vascular laboratory) plus symptoms of claudication; or
    - Amputation, peripheral bypass, or peripheral angioplasty of the extremities secondary to ischemia occurring at least 3 months (90 days) prior to the Screening visit (V1).

## Blinded data sample based in AVD CRF:

Table 14.1.2.11 (Ertugliflozin Protocol MK-8835-004/B1521021)
Subject Characteristics: Baseline CV Risk Factors, Diabetes Characteristics and Other Factors
CV ITT

| | Pla | (%) | Ertuglifl | (%) mg | Ertugliflo | zin 15 mg<br>(%) | All Erts | gliflozin<br>(%) | n Te | otal<br>(%) |
|---|---|---|---|---|---|---|---|---|---|---|
| Subjects in population | 2754 | | 2783 | | 2709 | | 5492 | | 8246 | |
| Albuninuria (mg/g) | i i | | | | 1 | | | | | |
| Normal-albuminuria (<30) | 1592 | (57.8) | 1587 | (57.0) | 1584 | (58.5) | 3171 | (57.7) | 4763 | (57.1 |
| Micro-albuminuria (≥30 to ≤300) | 820 | (29.8) | 870 | (31.3) | 796 | (29.4) | 1666 | (30.3) | 2486 | (30. |
| Macro-albuminuria (>300) | 268 | ( 9.7) | 242 | ( 3.7) | 244 | ( 9.0) | 486 | (8.8) | 754 | ( 9. |
| Unknown | 74 | (2.7) | 84 | ( 3.0) | 85 | ( 3.1) | 169 | ( 3.1) | 243 | ( 2 |
| History of Hypertension | | | | Y. | 1 | | | | | |
| No | 230 | ( 8.4) | 253 | ( 9.1) | 242 | ( 8.9) | 495 | ( 9.0) | 725 | ( 8. |
| Yes | 2524 | (91.6) | 2530 | (90.9) | 2467 | (91.1) | 4997 | (91.0) | 7521 | (91. |
| History of Dyslipidemia | | | 1 8 | 1 | | | | | | |
| No | 686 | (24.9) | 703 | (25.3) | 680 | (25.1) | 1383 | (25.2) | 2069 | (25. |
| Yes | 2068 | (75.1) | 2080 | (74.7) | 2029 | (74.9) | 4109 | (74.8) | 6177 | (74. |
| History of Coronary Artery Disease | | 1 | | | | | | | | |
| No | 680 | (24.7) | 670 | (24.1) | 640 | (23.6) | 1310 | (23.9) | 1990 | (24. |
| Yes | 2074 | (75.3) | 2113 | (75.9) | 2069 | (76.4) | 4182 | (76.1) | 6256 | (75. |
| History of Cerebrovascular Disease | | | | | | | | | | |
| No | 2135 | (77.5) | 2126 | (76.4) | 2094 | (77.3) | 4220 | (76.8) | 6355 | (77. |
| Yes | 619 | (22.5) | 657 | (23.6) | 615 | (22.7) | 1272 | (23.2) | 1891 | (22 |
| History of Peripheral Artery Disease | Par. | | | | | | | | | |
| No | 2199 | (79.8) | 2290 | (82.3) | 2215 | (81.8) | 4505 | (82.0) | 6704 | (81 |
| Yes | 555 | (20.2) | 493 | (17.7) | 494 | (18.2) | 987 | (18.0) | 1542 | (18 |

Data in Background publication - presented based on Medical History Blinded data:

Table 14.2.12.12.1 (Ertugliflozin Protocol MK-8835-004/B1521021) Selected Baseline CV Conditions CV ITT

| | Pla | cebo | Ertuglif | lozin 5 mg | Ertuglifle | ozin 15 mg | All Ertugliflozin | | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | п | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Subjects in population | 2754 | | 2783 | | 2709 | | 5492 | | 8246 | |
| Established CV disease | | | | 1 | P | | | | | |
| No | 19 | ( 0.7) | 22 | (0.8) | 18 | ( 0.7) | 40 | ( 0.7) | 59 | ( 0. |
| Yes | 2735 | (99.3) | 2761 | (99.2) | 2690 | (99.3) | 5451 | (99.3) | 8186 | (99. |
| MI (Cardiac SOC) | 1293 | (46.9) | 1346 | (48.4) | 1315 | (48.5) | 2661 | (48.5) | 3954 | (48. |
| Acute myocardial infarction | 222 | ( 8.1) | 236 | ( 8.5) | 224 | (8.3) | 460 | ( 8.4) | 682 | ( 8. |
| Myocardial infarction | 1084 | (39.4) | 1117 | (40.1) | 1103 | (40.7) | 2220 | (40.4) | 3304 | (40. |
| Silent myocardial infarction | 5 | ( 0.2) | 10 | ( 0.4) | 9 | ( 0.3) | 19 | ( 0.3) | 24 | ( 0. |
| Coronary revascularization (Procedures SOC) | 1598 | (58.0) | 1587 | (57.0) | 1605 | (59.2) | 3192 | (58.1) | 4790 | (58. |
| CABG | 602 | (21.9) | 621 | (22.3) | 592 | (21.9) | 1213 | (22.1) | 1815 | (22. |
| PCI | 1162 | (.42.2) | 1151 | (41.4) | 1176 | (43.4) | 2327 | (42.4) | 3489 | (42. |
| Coronary angioplasty | 273 | (9,9) | 292 | (10.5) | 266 | ( 9.8) | 558 | (10.2) | 831 | (10. |
| Coronary arterial stent insertion | 491 | (17.8) | 461 | (16.6) | 514 | (19.0) | 975 | (17.8) | 1466 | (17. |
| Coronary endarterectomy | 0 | ( 0.0) | 0 | (0.0) | 1 | ( 0.0) | 1 | ( 0.0) | 1 | ( 0.0 |
| Coronary revascularisation | 56 | ( 2.0) | 57 | ( 2.0) | 69 | ( 2.5) | 126 | ( 2.3) | 182 | ( 2. |
| Percutaneous coronary intervention | 471 | (17.1) | 493 | (17.7) | 485 | (17.9) | 978 | (17.8) | 1449 | (17.6 |
| Other | 61 | ( 2.2) | 61 | ( 2.2) | 74 | ( 2.7) | 135 | ( 2.5) | 196 | ( 2, |
| Stroke (Nervous system disorders) | 562 | (20.4) | 615 | (22.1) | 562 | (20.7) | 1177 | (21.4) | 1739 | (21. |
| Brain stem infarction | 0 | ( 0.0) | 4 | ( 0.1) | 1 | ( 0.0) | 5 | ( 0.1) | 5 | ( 0. |
| Brain stem stroke | 0 | ( 0.0) | 2 | ( 0.1) | 1 | ( 0.0) | 3 | ( 0.1) | 3 | ( 0.0 |

## $\label{eq:heaviside} \begin{aligned} & HF\ population\ \text{--}\ defined\ based\ on\ medical\ history\ \text{--}\ presented\ based\ on\ narrow\ Cardiac\ Failure\ SMQ \end{aligned}$

Table 14.2.12.12.1 (Ertugliflozin Protocol MK-8835-004/B1521021)
Selected Baseline CV Conditions
CV ITT

| | Pla | acebo | Ertuglif | lozin 5 mg | Ertuglifle | ozin 15 mg | All Ertugliflozin | | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Cerebellar infarction | 1 | ( 0.0) | 3 | ( 0.1) | _ 4 | ( 0.1) | 7 | ( 0.1) | 8 | ( 0.1) |
| Cerebral infarction | 24 | ( 0.9) | 32 | (1.1) | 31 | (1.1) | 63 | (1.1) | 87 | (1.1) |
| Cerebrovascular accident | 60 | ( 2.2) | 59 | (21) | 64 | ( 2.4) | 123 | ( 2.2) | 183 | ( 2.2) |
| Ischaemic cerebral infarction | 2 | ( 0.1) | 4 | ( 0.1) | 3 | ( 0.1) | 7 | ( 0.1) | 9 | ( 0.1) |
| Ischaemic stroke | 486 | (17.6) | 531 | (19.1) | 471 | (17.4) | 1002 | (18.2) | 1488 | (18.0) |
| Lacunar infarction | 9 | ( 0.3) | 9 | ( 0.3) | 5 | ( 0.2) | 14 | ( 0.3) | 23 | ( 0.3) |
| Thalamic infarction | 2 | ( 0.1) | 0 | ( 0.0) | 0 | ( 0.0) | 0 | ( 0.0) | 2 | ( 0.0) |
| Heart Failure | 654 | (23.7) | 652 | (23.4) | 627 | (23.1) | 1279 | (23.3) | 1933 | (23.4 |
| Acute left ventricular failure | 1 | ( 0.0) | 2 | ( 0.1) | 0 | ( 0.0) | 2 | ( 0.0) | 3 | ( 0.0 |
| Acute pulmonary oedema | 2 | (0.1) | 4.4 | ( 0.1) | 1 | ( 0.0) | 5 | ( 0.1) | 7 | ( 0.1 |
| Cardiac asthma | 0 | ( 0.0) | 1 | ( 0.0) | 2 | ( 0.1) | 3 | ( 0.1) | 3 | ( 0.0 |
| Cardiac failure | 9 🗐 | ( 0.3) | 8 | ( 0.3) | 14 | ( 0.5) | 22 | ( 0.4) | 31 | ( 0.4 |
| Cardiac failure acute | 0 | ( 0.0) | 0 | ( 0.0) | 1 | ( 0.0) | 1 | (0.0) | 1 | ( 0.0 |
| Cardiac failure chronic | 630 | (22.9) | 631 | (22.7) | 593 | (21.9) | 1224 | (22.3) | 1854 | (22.5 |
| Cardiac failure congestive | 8 | ( 0.3) | 7 | ( 0.3) | 5 | ( 0.2) | 12 | ( 0.2) | 20 | ( 0.2 |
| Cardiogenic shock | 1 | ( 0.0) | 0 | (0.0) | 0 | ( 0.0) | 0 | ( 0.0) | 1 | ( 0.0 |
| Chronic left ventricular failure | 0 | ( 0.0) | 1 | ( 0.0) | 0 | ( 0.0) | 1 | ( 0.0) | 1 | ( 0.0 |
| Cor pulmonale | 0 | ( 0.0) | 0 | (0.0) | 1 | ( 0.0) | 1 | ( 0.0) | 1 | ( 0.0 |
| Cor pulmonale chronic | 0 | ( 0.0) | 1 | ( 0.0) | 0 | ( 0.0) | 1 | (0.0) | 1 | ( 0.0 |
| Ejection fraction decreased | D 1 | ( 0.0) | 0 | ( 0.0) | 1 | ( 0.0) | 1 | ( 0.0) | 2 | ( 0.0 |
| Left ventricular failure | 8 | ( 0.3) | 7 | ( 0.3) | 12 | ( 0.4) | 19 | ( 0.3) | 27 | ( 0.3 |
| Pulmonary oedema | 6 | ( 0.2) | 6 | ( 0.2) | 7 | ( 0.3) | 13 | ( 0.2) | 19 | ( 0.2 |
| Ventricular faihure | 1 | ( 0.0) | 0 | ( 0.0) | 0 | ( 0.0) | 0 | ( 0.0) | 1 | ( 0.0 |


## NYHA – collected in subjects with HF at baseline – data collected retrospectively:

Table 14.2.12.12.1 (Ertugliflozin Protocol MK-8835-004/B1521021) Selected Baseline CV Conditions CV ITT

| | Pla | Placebo | | Ertugliflozin 5 mg | | Ertugliflozin 15 mg | | All Entugliflozin | | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | n | (%) | n | (%) | п | (%) | n | (%) | п | (%) |
| NYHA Functional Classification | | | | 0 | - | | | | | |
| Class I | 157 | ( 5.7) | 149 | (54) | 155 | ( 5.7) | 304 | ( 5.5) | 461 | ( 5.6 |
| Class II | 436 | (15.8) | 448 | (16.1) | 407 | (15.0) | 855 | (15.6) | 1291 | (15.7 |
| Class III | 50 | (1.8) | 49 | ( 1.8) | 44 | ( 1.6) | 93 | ( 1.7) | 143 | ( 1.7 |
| Class IV | 1 | ( 0.0) | 1.00 | ( 0.0) | 91 | ( 0.0) | 2 | ( 0.0) | 3 | ( 0.0 |
| Every subject is counted a single time for each applicable<br>bolded category. | specific condition. A subject | with multiple | e condition | within a bol | ded category | is counted a | single time | for that | | |
| Data cut date: 14Oct2019 | | | - 3 | ~ | | | | | | |
| PFIZER CONFIDENTIAL Date of Reporting Dataset Cr | estion: 12DEC2019 Date of | Table Cresti | on: 00IAN | 020(8:46) | | | | | | |

Source: [P004MK8835: adam-adsl; adcf; admh]

EF collection: data collection in all subjects if available. In case of multiple historical measurements in the same patient, sites were asked to repost EF based on the test obtained closest to randomization (prior to):

Table 14.2.12.15 (Ertugliflozin Protocol MK-8835-004/B1521021)

Classification of Ejection Fraction Prior to Randomization

CV ITT

| | Pia | cebo | Ertuglif | lozin 5 mg | Ertuglifle | ozin 15 mg | All Ertt | gliflozin | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | a | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Subjects in Population | 2754 | | 2783 | 3020 | 2709 | 11000 | 5492 | | 8246 | Artin |
| In the full CV ITT population | | | | 0 | Tool or | 10 | | | | |
| Subjects with EF data prior to randomization | 1678 | (60.9) | 1685 | (60.5) | 1642 | (60.6) | 3327 | (60.6) | 5005 | ( 60. |
| 0-1 year prior to randomization | 582 | (21.1) | 602 | (21.6) | 593 | (21.9) | 1195 | (21.8) | 1777 | (21. |
| EF reduced: ≤ 40% | 69 | ( 2.5) | 57 | ( 2.0) | 73 | ( 2.7) | 130 | (2.4) | 199 | ( 2 |
| EF preserved: > 40% | 513 | (18.6) | 545 | (19.6) | 520 | (19.2) | 1065 | (19.4) | 1578 | (19. |
| 0-2 year prior to randomization | 915 | (33.2) | 901 | (32.4) | 851 | (31.4) | 1752 | (31.9) | 2667 | (32. |
| EF reduced: ≤ 40% | 104 | (3.8) | 96 | ( 3.4) | 99 | ( 3.7) | 195 | ( 3.6) | 299 | ( 3. |
| EF preserved: > 40% | 811 | (29.4) | 805 | (28.9) | 752 | (27.8) | 1557 | (28.4) | 2368 | (28. |
| 0-3 year prior to randomization | 1105 | (40.1) | 1086 | (39.0) | 1046 | (38.6) | 2132 | (38.8) | 3237 | (39. |
| EF reduced: ≤ 40% | 123 | (4.5) | 122 | ( 4.4) | 125 | ( 4.6) | 247 | ( 4.5) | 370 | ( 4. |
| EF preserved: > 40% | 982 | (35.7) | 964 | (34.6) | 921 | (34.0) | 1885 | (34.3) | 2867 | (34. |
| 0-5 year prior to randomization | 1347 | (48.9) | 1335 | (48.0) | 1263 | (46.6) | 2598 | (47.3) | 3945 | (47. |
| EF reduced: ≤40% | 151 | ( 5.5) | 152 | ( 5.5) | 149 | ( 5.5) | 301 | ( 5.5) | 452 | ( 5. |
| EF preserved: > 40% | 1196 | (43.4) | 1183 | (42.5) | 1114 | (41.1) | 2297 | (41.8) | 3493 | (42. |
| Any time prior to randomization | 1678 | (60.9) | 1685 | (60.5) | 1642 | (60.6) | 3327 | (60.6) | 5005 | (60. |
| EF reduced: ≤ 40% | 179 | ( 6.5) | 173 | ( 6.2) | 189 | ( 7.0) | 362 | ( 6.6) | 541 | ( 6. |
| EF preserved: > 40% | 1499 | (54.4) | 1512 | (54.3) | 1453 | (53.6) | 2965 | (54.0) | 4464 | (54. |

Table 14.2.12.15 (Ertugliflozin Protocol MK-8835-004/B1521021)

Classification of Ejection Fraction Prior to Randomization

CV ITT

| | Pts | Placebo | | lozin 5 mg | Ertuglifle | ozin 15 mg | All Em | ugliflozin | T | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| In subjects with a history of heart failure | | | | - | Diam. | | | | | |
| Subjects with EF data prior to randomization 2 | 498 | | 492 | - 0 | 476 | | 968 | | 1466 | |
| 0-1 year prior to randomization | 204 | (41.0) | 208 | (42.3) | 211 | (44.3) | 419 | (43.3) | 623 | (42.5) |
| EF reduced: ≤ 40% | 42 | ( 8.4) | 37 | ( 7.5) | 46 | ( 9.7) | 83 | ( 8.6) | 125 | ( 8.5) |
| EF preserved: > 40% | 162 | (32.5) | 171 | (34,8) | 165 | (34.7) | 336 | (34.7) | 498 | (34.0) |
| 0-2 year prior to randomization | 319 | (64.1) | 312 | (63.4) | 289 | (60.7) | 601 | (62.1) | 920 | (62.8) |
| EF reduced: ≤ 40% | 61 | (12.2) | 63 | (12.8) | 60 | (12.6) | 123 | (12.7) | 184 | (12.6) |
| EF preserved: > 40% | 258 | (51.8) | 249 | (50.6) | 229 | (48.1) | 478 | (49.4) | 736 | (50.2) |
| 0-3 year prior to randomization | 359 | (72.1) | 362 | (73.6) | 338 | (71.0) | 700 | (72.3) | 1059 | (72.2) |
| EF reduced: ≤ 40% | 70 | (141) | 71 | (14.4) | 73 | (15.3) | 144 | (14.9) | 214 | (14.6) |
| EF preserved: > 40% | 289 | (58.0) | 291 | (59.1) | 265 | (55.7) | 556 | (57.4) | 845 | (57.6) |
| 0-5 year prior to randomization | 433 | (86.9) | 419 | (85.2) | 392 | (82.4) | 811 | (83.8) | 1244 | (84.9) |
| EF reduced: ≤ 40% | 81 | (16.3) | 83 | (16.9) | 86 | (18.1) | 169 | (17.5) | 250 | (17.1) |
| EF preserved: > 40% | 352 | (70.7) | 336 | (68.3) | 306 | (64.3) | 642 | (66.3) | 994 | (67.8) |
| Any time prior to randomization | 498 | (100.0) | 492 | (100.0) | 476 | (100.0) | 968 | (100.0) | 1466 | (100.0 |
| EF reduced: ≤ 40% | 93 | (18.7) | 91 | (18.5) | 99 | (20.8) | 190 | (19.6) | 283 | (19.3) |
| EF preserved: > 40% | 405 | (813) | 401 | (81.5) | 377 | (79.2) | 778 | (80.4) | 1183 | (80.7) |

Subjects with FE data are classified in all applicable time periods based on the most recent FF results prior to randomization.

History of heart failure is defined as baseline condition coding to manow heart failure SMQ.

Data cut date: 14Oct2019

PFIZER CONFIDENTIAL Date of Reporting Dataset Creation: 08JAN2020 Date of Table Creation: 08JAN2020(17:48)

Source: [P004MK8835: adam-adsl; adbase]

## Reference points from publications:


<sup>1</sup> Used as the denominator for all categories below.

EF = ejection fraction.

## DAPA HF-NEJM (contribution of urgent visits was minimal to overall endpoints pool)

| Variable | Dapag<br>(N= | liflozin<br>2373) | Plac<br>(N=3 | | Hazard or Rate Ratio<br>or Difference<br>(95% CI) | P Value |
|---|---|---|---|---|---|---|
| | values | events/100<br>patient-yr | values | events/100<br>patient-yr | | |
| Efficacy outcomes | | | | | | |
| Primary composite outcome — no. (%)† | 386 (16.3) | 11.6 | 502 (21.2) | 15.6 | 0.74 (0.65 to 0.85) | < 0.001 |
| Hospitalization or an urgent visit for heart failure | 237 (10.0) | 7.1 | 326 (13.7) | 10.1 | 0.70 (0.59 to 0.83) | NA |
| Hospitalization for heart failure | 231 (9.7) | 6.9 | 318 (13.4) | 9.8 | 0.70 (0.59 to 0.83) | NA |
| Urgent heart-failure visit | 10 (0.4) | 0.3 | 23 (1.0) | 0.7 | 0.43 (0.20 to 0.90) | NA |
| Cardiovascular death | 227 (9.6) | 6.5 | 273 (11.5) | 7.9 | 0.82 (0.69 to 0.98) | NA |